CLINICAL TRIAL: NCT05495620
Title: Real-world Evidence of Carfilzomib, Lenalidomide, Dexamethasone Combination Therapy in Korean Relapsed and/or Refractory Multiple Myeloma Patients
Brief Title: Long-term KRd in Relapsed and/or Refractory Multiple Myeloma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Dong-A University Hospital (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Sung-Hyun Kim, Professor, Dong-A University Hospital
Other Study IDs: DAUHIRB-22-081
Record Dates: First submitted 2022-07-05; First posted 2022-08-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Multiple Myeloma in Relapse; Multiple Myeloma, Refractory
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Relapsed and/or refractory multiple myeloma: Multiple myeloma in relapsed but not refractory, relapsed and refractory, and primary refractory status
  Interventions: Drug: Carfilzomib; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib — Intravenous
  carfilzomib, lenalidomide, dexamethasone
  Other Names: Kyprolis
Drug: Lenalidomide — Oral
  Other Names: Revlimid
Drug: Dexamethasone — Oral or intravenous

SUMMARY:
Research question: Is KRd therapy effective and safe in the real-world Asian patients?

Primay objective: To evaluate the effectiveness of KRd in RRMM patients

Secondary objectives:

To evaluate the effectiveness of investigational treatment strategy by

* PFS difference according to the high-risk disease subgroups and previous treatment
* OS
* Overall response rate and clinical benefit rate
* Duration of response To evaluate the safety and tolerability of KRd in RRMM patients

DETAILED DESCRIPTION:
Key study variables:

Demographic data, ISS, R-ISS, cytogenetic abnormalities on FISH and G-banding, previous treatment regimens, response to previous treatment regimens, existence of extramedullary plasmacytoma, MM-related symptoms, whether or not M protein has increased twice or more in 2-3 months at the time of KRd commencement, response to KRd therapy, duration of KRd treatment, adverse events during KRd therapy, disease progression and progression date, survival, and censored date or day of death

ELIGIBILITY:
Inclusion criteria

1. Patients ≥ 19 years
2. Relapsed and/or refractory multiple myeloma patients
3. Patients who had received KRd combination chemotherapy from February, 2018 to February, 2020.

Exclusion criteria

1. Patient who had not been treated with KRd combination therapy from the first cycle of treatment
2. Patients who had received KRd combination chemotherapy before February, 2018 and after February, 2020.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Relapsed and/or refractory multiple myeloma patients treated with carfilzomib-lenalidomide-dexamethasone combination chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | up to 54 months
  the time from the first date of KRd to the date of disease progression or death or censored date

SECONDARY OUTCOMES:
Overall survival | up to 54 months
  the time from the first date of KRd treatment to the time of death or censored date
Overall response rate, clinical benefit rate | up to 54 months
  the proportion of patients who achieved a PR or better, which response is defined by the IMWG criteria, the proportion of patients who achieved a MR or better
Duration of response | up to 54 months
  the time from the first date of response to the time of disease progression or death or censored date
Toxicity profile | up to 2 years
  toxicities as determined by the incidence of clinical and laboratory findings occurred from the time of the first date of KRd treatment to the date of disease progression or death or censored date

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Hyun Kim, MD, Ph.D, Principal Investigator — Dong-A University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stewart AK, Rajkumar SV, Dimopoulos MA, Masszi T, Spicka I, Oriol A, Hajek R, Rosinol L, Siegel DS, Mihaylov GG, Goranova-Marinova V, Rajnics P, Suvorov A, Niesvizky R, Jakubowiak AJ, San-Miguel JF, Ludwig H, Wang M, Maisnar V, Minarik J, Bensinger WI, Mateos MV, Ben-Yehuda D, Kukreti V, Zojwalla N, Tonda ME, Yang X, Xing B, Moreau P, Palumbo A; ASPIRE Investigators. Carfilzomib, lenalidomide, and dexamethasone for relapsed multiple myeloma. N Engl J Med. 2015 Jan 8;372(2):142-52. doi: 10.1056/NEJMoa1411321. Epub 2014 Dec 6. PMID 25482145